CLINICAL TRIAL: NCT04008667
Title: The Effect of Acupoint Application on Postoperative Ileus: a Randomized Controlled Trial
Brief Title: The Effect of Acupoint Application on Postoperative Ileus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: li xiong (Other)
Responsible Party: Sponsor-Investigator, li xiong, Professor, Central South University
Organization: Central South University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: lxiong
Record Dates: First submitted 2019-06-29; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Postoperative Ileus
Keywords: Postoperative ileus; acupoint; ERAS; Chinese medicine

STUDY DESIGN:
Intervention Model Description: Intervention arm：receiving acupoint application and regular therapy; Placebo arm: receiving fake acupoint application and regular therapy; control arm: receiving regular therapy.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention arm (Experimental): Receiving the acupoint application and optimal supports.
  The patients start using the acupoint application on the umbilical Shenque point in 2 hours after surgery, 1 or 2 times a day, lasting 5 days.
  All patients will receive optimal supports during the observation period, including preoperative gastrointestinal preparation, inserting gastric tube, postoperative fasting, necessary antibiotic use, rational fluid management, detaining drainage tube, etc.
  Interventions: Other: Acupoint application
- Placebo arm (Placebo Comparator): Receiving the fake acupoint application and optimal supports.
  The fake acupoint is
  The patients start using the fake acupoint application on the umbilical Shenque point in 2 hours after surgery, 1 or 2 times a day, lasting 5 days.
  All patients will receive optimal supports during the observation period, including preoperative gastrointestinal preparation, inserting gastric tube, postoperative fasting, necessary antibiotic use, rational fluid management, detaining drainage tube, etc.
  Interventions: Other: Fake acupoint application
- Control arm (No Intervention): Receiving the optimal supports.
  All patients will receive optimal supports during the observation period, including preoperative gastrointestinal preparation, inserting gastric tube, postoperative fasting, necessary antibiotic use, rational fluid management, detaining drainage tube, etc.

INTERVENTIONS:
Other: Acupoint application — Acupoint application: The patients start using the acupoint application on the umbilical Shenque point in 2 hours after surgery, 1 or 2 times a day, lasting 5 days.
  Arms: Intervention arm
Other: Fake acupoint application — Fake acupoint application: The patients start using the fake acupoint application on the umbilical Shenque point in 2 hours after surgery, 1 or 2 times a day, lasting 5 days.
  Arms: Placebo arm

SUMMARY:
This study aims to verify the therapeutical effect and mechanism of acupoint application on postoperative ileus.

DETAILED DESCRIPTION:
Postoperative ileus (POI) is a common disorder of gastrointestinal motility characterized by abdominal distension, nausea, vomiting and delayed passage of flatus or stool, which develops after every abdominal surgical procedure. POI increases risk of developing postoperative complications, decreases the bed turnover rate and prolongs the average duration of hospitalization, increasing the expense of both patients and hospitals. Although the Pathophysiological mechanism of POI remains unclear, recent researches suggests the inflammatory responses after surgery might be responsible for the gastrointestinal motility disorder. Acupoint application is a traditional chinese intervention which has been used in treating gastrointestinal motility disorder resulted from other causes. In this study, we aims to verify the therapeutical effect and mechanism of acupoint application on postoperative ileus.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients are scheduled to undergo elective abdominal surgery;
* 2. Patients age between 20 to 80 years old;
* 3. Umbilical skin condition is good;
* 4. Written informed consent provided to participate in the study.

Exclusion Criteria:

* 1.Patients don't match the inclusion criteria;
* 2. Patients with severe comorbidity such as cardiac disease, liver disease, pulmonary disease or renal disease ;
* 3.Patients with mental disorder;
* 4. Patients have gastrointestinal mobility disorder resulted from clear causes, such as ankylenteron, ascites, etc;
* 5. Patients received ostomy operation, such as jejunostomy;
* 6.Patients who have history of abdominal surgery or history of bowel obstruction;
* 7. Patients who receive other treatments to improve the gastrointestinal mobility or/and to relieve POI related symptoms , such as gastrointestinal prokinetic drugs, enema, etc.
* 8. Patients who are allergic to the acupoint applicaton;
* 9.Patients who are unsuitable for study inclusion as determined by the investigator. (eg: patients with severe operation related complications)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2019-07 (Estimated); Primary Completion 2021-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
time to defecate and tolerate for food (TF+D) | End of surgery to time to defecate and tolerate for food(from 5 to 7 days)
  Defined as the first time that the patient could both defecate and tolerate orally taking food after surgery.

SECONDARY OUTCOMES:
time to return of bowel sounds | End of surgery to the first bowel sound (from 1 to 5 days)
  Defined as the first time hear the bowel sound after surgery.
time to report of first flatus | End of surgery to the first flatus (from 1 to 5 days)
  Defined as the first time flatus happens.
time to report of first defecation | End of surgery to the first defecation. (from 1 to 7 days)
  Defined as the first time defecation happens.
length of postoperative hospitalization | End of surgery to hospital discharge. (from 5 to 7 days)
  Defined as the length hospitalization after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No